Chronic postsurgical pediatric pain. Observational Study. Guillermo Ceniza-Bordallo et al. 15 December 2020. University Complutense of Madrid.





## CHRONIC POSTSURGICAL PEDIATRIC PAIN.

**TITLE:** RISK FACTORS TO DEVELOP CHRONIC POSTSURGICAL PEDIATRIC PAIN

**INVESTIGATOR PRINCIPAL:** GUILLERMO CENIZA-BORDALLO

**PROJECT ENTITIES:** COMPLUTENSE UNIVERSITY OF MADRID & 12 OCTUBRE PEDIATRIC HOSPITAL.

**NUMBER OF IDENTIFIACTION: 26/618** 

**DATE:** 15<sup>TH</sup> December 2020.

Chronic postsurgical pediatric pain. Observational Study. Guillermo Ceniza-Bordallo et al. 15 December 2020. University Complutense of Madrid.





## **Statistical Analysis Plan**

The results will be analyzed with the SPSS 25 statistical program (SPSS, Inc., Chicag0, IL, USA). The interpretation of the statistical tests will be carried out based on a significance level of 5% (P <0.05). First, the demographic variables of the sample will be presented as mean  $\pm$  standard deviation (SD), in the case of quantitative variables, and as an absolute value (relative frequency percentage in the case of qualitative variables).

The correlation of the risk factors of both children and parents with chronic post-surgical pain in children will be analyzed. To do this, the Pearson Correlation Coefficient will be used, categorizing the magnitude of the correlation as follows: strong (> 0.60), moderate (0.30-0.60), and weak or very weak (<0.30).

Additionally, a multiple linear regression model will be used to determine the degree of association between risk factors and chronic postsurgical pain. Specifically, the intensity and location of pain will be included as criterion variables, while catastrophizing, anxiety, fear of pain, fear of movement and quality of life will be considered as predictor variables. The degree of multicollinearity existing between the predictor variables will be evaluated using the Variance Inflation Factor (VIF). The strength of association will be examined using the adjusted coefficient of determination (adjusted R2). In addition, the regression coefficient (B), the P-value and the standardized beta coefficient ( $\beta$ ) will be calculated for each predictor variable of the reduced final model. Thus, it will be possible to determine the variables that most directly influence the regression model.